CLINICAL TRIAL: NCT03191487
Title: Evaluation of a New Organization for Collecting Pre-chemotherapy Session Information: a Multicenter, Open, Randomized Trial
Brief Title: Evaluation of a New Organization for Collecting Pre-chemotherapy Session Information
Acronym: ChimioPal
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no Financial agreement
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PREPS/2016/MF-01
Record Dates: First submitted 2017-06-15; First posted 2017-06-19 (Actual); Last update posted 2017-06-19 (Actual); Status verified 2017-06

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ChimioPal (Experimental): Systematic collection of clinical and laboratory toxicities.
  Interventions: Other: ChimioPal
- Standard (Active Comparator): The usual management and logistic pathways will be respected.
  Interventions: Other: Usual pathways

INTERVENTIONS:
Other: ChimioPal — Systematic collection of clinical and laboratory toxicities (TXs) during the 2-4 days preceding a chemotherapy (CT) session (48H before a session (D-2 towards the end of the afternoon) and a maximum of 96h before sessions occurring on Mondays (D-4 towards the end of the afternoon). Clinical TX data will be collected via ChimioPal (a self-questionnaire administered by smartphone) and laboratory TX data will be collected via Apicrpyt (secure messaging service) or a fax-to-email service. Data flow management by a nurse dedicated to this activity in each centre will be implemented. If the results of the assessment do not authorize CT, additional assessments may be prescribed. If the experimental data transmission does not occur, the usual pathways will be implemented.
  Patient training on how to use a smart phone and the questionnaire will be performed by a nurse before the start of the first chemotherapy session, with reminders at the following sessions if required.
  Arms: ChimioPal
Other: Usual pathways — In the standard arm, the usual management and logistic pathways will be respected. Only extra data collection is required by this study.
  Arms: Standard

SUMMARY:
The primary objective of this study is to compare an experimental organization for chemotherapy session planning based on early, standardized, and prioritized means of data transmission via secure e-mail (laboratory results) and the use of a smart phone (for clinical toxicity data) compared to the regular organization, in terms of the rate of prescriptions of chemotherapy prepared at the latest the day before a session and then administered in full (over a 6-month observation period) among colorectal cancer patients in need of cancer treatment in an outpatient setting.

DETAILED DESCRIPTION:
Compare the two arms of the study in terms of:

A. each element contributing to the primary criterium;

B. the quality of chemotherapy related care;

C. logistics;

D. patient satisfaction with respect to support for chemotherapy care;

E. the feasibility and acceptability of the organization by patients will be assessed by the rate of optimal use of toxicity collection tools and patient satisfaction rates relative to the tool (experimental arm)

F. Comparison of the overall cost of care in both arms and estimated cost of the strategy

ELIGIBILITY:
Inclusion Criteria:

* The patient was informed about the implementation of the study, its objectives, constraints and patient rights
* The patient has given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient is available for 6 months of follow-up
* The patient is treated via anti-cancer chemotherapy for colorectal cancer
* The patient is starting a new adjuvant or metastatic chemotherapy protocol with a follow-up in a day-clinic setting
* The patient has already used a smartphone, or desires to learn how, or is accompanied by a person who can help the patient use a smartphone
* The anticipated chemotherapy treatment corresponds to one of the following protocols: cetuximab, FOLFIRI, FOLFIRI-aflibercept, FOLFIRI-bevacizumab, FOLFIRI-cetuximab, FOLFIRI-panitumumab, Folfirinox, Folfirinox-bevacizumab, Folfoxiri, Folfoxiri-bevacizumab, FOLFOX 4 simplified, FOLFOX 4 simplified - bevacizumab, FOLFOX 4 simplified - cetuximab, FOLFOX 4 simplified - panitumumab, Irinotecan-cetuximab, LV5FU2 simplified, panitumumab, XELOX.

Exclusion Criteria:

* The patient is participating in another study, or has participated in another study within the past 3 months, that may influence the results or conclusions of the present trial
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, or is an adult under guardianship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient is pregnant, parturient, or breastfeeding
* The planned chemotherapy regimen includes weekly treatment cycles
* Patient who is incapable of using a smartphone either by himself/herself or via another helping person

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-04 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
The rate of prescriptions for chemotherapy in the outpatient clinic prepared at the latest the day before a session (except for predefined, limited stability products) and administered in full, per patient, during a follow-up period of 6 months | 6 months
  This criterion is aggregated per patient but its components are collected for each prescription, according to the following coding:
  * Prescription prepared in advance and administered in full: 1
  * Prescription prepared in advance but not administered in full: 0
  * Prescription not prepared in advance : 0
  For each patient, the sum of the results for each prescription will be the numerator. The denominator is the number of prescriptions during 6 months follow-up for each patient.
  The limited stability products that will necessarily be prepared at the last minute are:
  * Aflibercept
  * Panitumumab
  * Raltitrexed

SECONDARY OUTCOMES:
The number of prescriptions prepared in advance and administered in full | 6 months
The number of prescriptions prepared in advance and not administered in full | 6 months
The number of prescriptions not prepared in advance | 6 months
Dose-intensity per patient over 6 months of follow-up | 6 months
The number of chemotherapy session postponements that were anticipated, and the patient was not required to come in to the clinic | 6 months
The number of chemotherapy session postponements that were not anticipated, and the patient was required to come in to the clinic | 6 months
The number of pharmaceutical interventions* accepted by the doctor / the number of prescriptions prepared for the totality of sessions | 6 months
  *a pharmaceutical intervention = request for prescription verification following results/information
The number of chemotherapy sessions that really took place (c) during the 6 months of follow-up | 6 months
The average number of days between chemotherapy sessions | 6 months
  The average number of days of inter-session lag:
  ∑(days between 2 sessions-expected days between 2 sessions)/(c-1)
The waiting time (on average) for the patient in the outpatient clinic before administration of the treatment | 6 months
the total period of time spent by the patient in the outpatient clinic | 6 months
The number of prescriptions that were prepared and administered | 6 months
The number of pouches that were prepared, not-administered, but recycled | 6 months
The number of pouches prepared, not administered and destroyed | 6 months
The average number of laboratory assessments required per chemotherapy session | 6 months
Patient satisfaction vis-à-vis their chemotherapy care (Visual Analog Scale from 0.0 to 10.0) | 6 months
Experimental arm per patient: The number Apicrypt transmissions / number of lab prescriptions | 6 months
Experimental arm per patient: the number questionnaires filled out / the number of requested questionnaires | 6 months
Experimental arm: Patient satisfaction vis-à-vis the ChimioPal tool (Visual Analog Scale from 0.0 to 10.0) | 6 months
Overall costs | 6 months
  The cost of pouches, consultations, examinations and transport will be estimated in both arms. Staff time, optimized due to the new organization, will be quantified. The point of view of health insurance and the establishment will be considered. Any gains will be weighed against the cost of the experimental strategy.

CONTACTS AND LOCATIONS:
Overall Officials: Mireille Favier, PharmD, Study Director — Centre Hospitalier Universitaire de Nîmes
Locations (6):
- France (6):
  - Institut Sainte Catherine, Avignon
  - Institut de Cancérologie Montpellier, Montpellier
  - CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes
  - CHRU de Strasbourg - Hôpital de Hautepierre, Strasbourg
  - CHRU de Toulouse - Hôpital de Rangueil, Toulouse
  - IUCT-Oncopole, Toulouse